CLINICAL TRIAL: NCT02218203
Title: Clinical Neuropharmacology of Pain in Spinal Cord Injury- Dextromethorphan/Lidocaine Combination (Factorial Design) Clinical Trial
Brief Title: Clinical Neuropharmacology of Pain in Spinal Cord Injury- Dextromethorphan/Lidocaine Combination Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Christine N. Sang, MD, MPH, Director, Translational Pain Research, Brigham and Women's Hospital
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2000p001387; R01NS041503 (NIH)
Record Dates: First submitted 2014-08-13; First posted 2014-08-18 (Estimated); Results first posted 2018-03-22 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-11

CONDITIONS: Central Neuropathic Pain; Allodynia; Spinal Cord Injury
Keywords: chronic pain; central neuropathic pain; spinal cord injury; dextromethorphan; lidocaine; combination therapy; analgesia
MeSH Terms: conditions — Hyperalgesia; Spinal Cord Injuries; Chronic Pain; Agnosia | interventions — Dextromethorphan; Lidocaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (16):
- Placebo- 0mg/kg Lido (Placebo Comparator): Placebo in combination with 0mg/kg LBM lidocaine
  Interventions: Drug: Placebo (Dextromethorphan); Drug: Placebo (Lidocaine)
- Placebo - 1mg/kg Lido (Experimental): Placebo in combination with 1mg/kg LBM lidocaine
  Interventions: Drug: Lidocaine; Drug: Placebo (Dextromethorphan)
- Placebo - 2mg/kg Lido (Experimental): Placebo in combination with 2mg/kg LBM lidocaine
  Interventions: Drug: Lidocaine; Drug: Placebo (Dextromethorphan)
- Placebo - 4mg/kg Lido (Experimental): Placebo in combination with 4mg/kg LBM lidocaine
  Interventions: Drug: Lidocaine; Drug: Placebo (Dextromethorphan)
- Low Dose Dex - 0mg/kg Lido (Experimental): Low dose dextromethorphan in combination with 0mg/kg LBM lidocaine
  Interventions: Drug: Dextromethorphan; Drug: Placebo (Lidocaine)
- Low Dose Dex - 1mg/kg Lido (Experimental): Low dose dextromethorphan in combination with 1mg/kg LBM lidocaine
  Interventions: Drug: Dextromethorphan; Drug: Lidocaine
- Low Dose Dex - 2mg/kg Lido (Experimental): Low dose dextromethorphan in combination with 2mg/kg LBM lidocaine
  Interventions: Drug: Dextromethorphan; Drug: Lidocaine
- Low Dose Dex - 4mg/kg Lido (Experimental): Low dose dextromethorphan in combination with 4mg/kg LBM lidocaine
  Interventions: Drug: Dextromethorphan; Drug: Lidocaine
- Medium Dose Dex - 0mg/kg Lido (Experimental): Medium dose dextromethorphan in combination with 0mg/kg LBM lidocaine
  Interventions: Drug: Dextromethorphan; Drug: Placebo (Lidocaine)
- Medium Dose Dex - 1mg/kg Lido (Experimental): Medium dose dextromethorphan in combination with 1mg/kg LBM lidocaine
  Interventions: Drug: Dextromethorphan; Drug: Lidocaine
- Medium Dose Dex - 2mg/kg Lido (Experimental): Medium dose dextromethorphan in combination with 2mg/kg LBM lidocaine
  Interventions: Drug: Dextromethorphan; Drug: Lidocaine
- Medium Dose Dex - 4mg/kg Lido (Experimental): Medium dose dextromethorphan in combination with 4mg/kg LBM lidocaine
  Interventions: Drug: Dextromethorphan; Drug: Lidocaine
- High Dose Dex - 0mg/kg Lido (Experimental): High dose dextromethorphan in combination with 0mg/kg LBM lidocaine
  Interventions: Drug: Dextromethorphan; Drug: Placebo (Lidocaine)
- High Dose Dex - 1mg/kg Lido (Experimental): High dose dextromethorphan in combination with 1mg/kg LBM lidocaine
  Interventions: Drug: Dextromethorphan; Drug: Lidocaine
- High Dose Dex - 2mg/kg Lido (Experimental): High dose dextromethorphan in combination with 2mg/kg LBM lidocaine
  Interventions: Drug: Dextromethorphan; Drug: Lidocaine
- High Dose Dex - 4mg/kg Lido (Experimental): High dose dextromethorphan in combination with 4mg/kg LBM lidocaine
  Interventions: Drug: Dextromethorphan; Drug: Lidocaine

INTERVENTIONS:
Drug: Dextromethorphan — Administered in 4 periods (placebo, low dose, medium dose, and high dose) for each subject, relative to each subject's MTD)
  Arms: High Dose Dex - 0mg/kg Lido; High Dose Dex - 1mg/kg Lido; High Dose Dex - 2mg/kg Lido; High Dose Dex - 4mg/kg Lido; Low Dose Dex - 0mg/kg Lido; Low Dose Dex - 1mg/kg Lido; Low Dose Dex - 2mg/kg Lido; Low Dose Dex - 4mg/kg Lido; Medium Dose Dex - 0mg/kg Lido; Medium Dose Dex - 1mg/kg Lido; Medium Dose Dex - 2mg/kg Lido; Medium Dose Dex - 4mg/kg Lido
Drug: Lidocaine — 0mg, 1mg, 2mg, and 4mg Lidocaine per kg of lean body mass (LBM), during each of the 4 dextromethorphan periods (placebo, low dose, medium dose, and high dose)
  Arms: High Dose Dex - 1mg/kg Lido; High Dose Dex - 2mg/kg Lido; High Dose Dex - 4mg/kg Lido; Low Dose Dex - 1mg/kg Lido; Low Dose Dex - 2mg/kg Lido; Low Dose Dex - 4mg/kg Lido; Medium Dose Dex - 1mg/kg Lido; Medium Dose Dex - 2mg/kg Lido; Medium Dose Dex - 4mg/kg Lido; Placebo - 1mg/kg Lido; Placebo - 2mg/kg Lido; Placebo - 4mg/kg Lido
Drug: Placebo (Dextromethorphan) — 0mg Dextromethorphan
  Arms: Placebo - 1mg/kg Lido; Placebo - 2mg/kg Lido; Placebo - 4mg/kg Lido; Placebo- 0mg/kg Lido
Drug: Placebo (Lidocaine) — 0mg/kg LBM Lidocaine
  Arms: High Dose Dex - 0mg/kg Lido; Low Dose Dex - 0mg/kg Lido; Medium Dose Dex - 0mg/kg Lido; Placebo- 0mg/kg Lido

SUMMARY:
This randomized, placebo-controlled, double-blind 4x4 crossover clinical trial was part of a larger NIH-funded study to evaluate the analgesic efficacy of multiple dose-combinations of chronic oral (PO) dextromethorphan and intravenous (IV) lidocaine in central neuropathic pain following spinal cord injury.

DETAILED DESCRIPTION:
This trial has several objectives:

Primary Objective To determine which combination (dose-ratio) of dextromethorphan and lidocaine provides the best balance of pain reduction and toxicity.

Secondary Objectives include To evaluate the analgesic efficacy of both dextromethorphan and lidocaine in attenuating pain related to central nervous system sensitization, specifically spontaneous pain, mechanical allodynia, and hyperalgesia.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female adults, age 18 to 70 with central neuropathic pain for a minimum of 3 months following SCI as confirmed by neurologic evaluation, with an average pain intensity score of at least moderate over at least 50% of the day for the 7 days prior to the screening visit and over the 7 days prior to starting study medication.
2. Subjects used no medication or a stabilized medication regimen for chronic and well-controlled medical conditions
3. Serum laboratory examination obtained at study entry:
4. Normal cognitive function.
5. Signed informed consent.

Exclusion Criteria:

1. Pregnancy or breast-feeding.
2. Renal or hepatic dysfunction.
3. Significant cardiac disease (e.g. MI within 1 year).
4. Signs or symptoms of central neurological disorder, excluding SCI.
5. Severe psychological disorder requiring treatment.
6. History of hypersensitivity or intolerance to dextromethorphan or lidocaine.
7. Participation in a study of an investigational drug or device within 30 days prior to screening for this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2003-04; Primary Completion 2008-01 (Actual); Study Completion 2008-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Christine N. Sang, MD, MPH, Principal Investigator — Translational Pain Research, Brigham and Women's Hospital (Disclosure: Patent)
Locations (1):
- Translational Pain Research, Brigham and Women's Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Translational Pain Research, Brigham and Women's Hospital — http://www.paintrials.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in March 2003. Subjects were recruited nationally from referring physicians, through advertisements, and through an existing database held by the PI.
Pre-assignment Details: During the screening visit, P450 2D6 phenotype status was determined for each subject to identify dextromethorphan-metabolizing capacity; those who were P450 2D6 poor-metabolizers were excluded. Following screen, subjects entered a dose escalation study to determine their maximum tolerated dose of dextromethorphan, prior to randomization.
Groups:
- Dextromethorphan/Lidocaine Combination Clinical Trial: This randomized, placebo-controlled, double-blind 4x4 factorial crossover clinical trial was part of a larger NIH-funded study to evaluate the analgesic efficacy of multiple dose-combinations of chronic oral (PO)dextromethorphan (placebo, low dose, medium dose, and high dose) and intravenous (IV) lidocaine (0mg/kg LBM, 1mg/kg LBM, 2mg/kg LBM, and 4mg/kg LBM) in central neuropathic pain following spinal cord injury.
Period: Overall Study
Arm/Group | Dextromethorphan/Lidocaine Combination Clinical Trial
Started | 26
Placebo Dex v. 0mg/km LBM Lidocaine | 24
Placebo Dex v. 1mg/km LBM Lidocaine | 24
Placebo Dex v. 2mg/km LBM Lidocaine | 24
Placebo Dex v. 4mg/km LBM Lidocaine | 24
Low Dose Dex v. 0mg/km LBM Lidocaine | 26
Low Dose Dex v. 1mg/km LBM Lidocaine | 26
Low Dose Dex v. 2mg/km LBM Lidocaine | 26
Low Dose Dex v. 4mg/km LBM Lidocaine | 26
Medium Dose Dex v. 0mg/km LBM Lidocaine | 24
Medium Dose Dex v. 1mg/km LBM Lidocaine | 24
Medium Dose Dex v. 2mg/km LBM Lidocaine | 24
Medium Dose Dex v. 4mg/km LBM Lidocaine | 24
High Dose Dex v. 0mg/km LBM Lidocaine | 24
High Dose Dex v. 1mg/km LBM Lidocaine | 24
High Dose Dex v. 2mg/km LBM Lidocaine | 24
High Dose Dex v. 4mg/km LBM Lidocaine | 24
Completed | 26 (2 subjects did not complete the placebo, medium dose, and high dose dex/lido combination arms.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Dextromethorphan/Lidocaine Combination Clinical Trial
Number analyzed (Participants) | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 25
  >=65 years | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 46.84 (11.32)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14
  Male | 12
Region of Enrollment [Number; unit: participants]
  North America | 26

OUTCOME MEASURES:

1. Primary Outcome: Percent Change in Peak Pain Intensity
Description: Primary outcome was percent change from baseline in mean pain intensity at Cmax (transformed Gracely Scale; 0-35). Higher values on the Gracely scale represent greater pain intensity; the greater the percent change from baseline in mean pain intensity, the bigger the reduction in pain intensity.
Time Frame: 30 minutes post-infusion (Cmax)
Population: Central neuropathic pain following SCI; we present the primary efficacy endpoint (percent change in peak pain intensity) of this nested IV lidocaine dose-response clinical trial independent of the dextromethorphan doses, because the distribution of the dextromethorphan doses is balanced across the lidocaine treatment arms.
Measure: Mean (Standard Error); unit: percentage change from baseline
Groups:
- Dextromethorphan/ 0mg/kg Lidocaine Combination: This randomized, placebo-controlled, double-blind 4x4 factorial crossover clinical trial was part of a larger NIH-funded study to evaluate the analgesic efficacy of multiple dose-combinations of chronic oral (PO)dextromethorphan (placebo, low dose, medium dose, and high dose) and intravenous (IV) lidocaine (0mg/kg LBM, 1mg/kg LBM, 2mg/kg LBM, and 4mg/kg LBM) in central neuropathic pain following spinal cord injury. This arm represents an average of all dextromethorphan doses in combination with 0mg/kg Lidocaine.
- Dextromethorphan/1mg/kg Lidocaine Combination: This randomized, placebo-controlled, double-blind 4x4 factorial crossover clinical trial was part of a larger NIH-funded study to evaluate the analgesic efficacy of multiple dose-combinations of chronic oral (PO)dextromethorphan (placebo, low dose, medium dose, and high dose) and intravenous (IV) lidocaine (0mg/kg LBM, 1mg/kg LBM, 2mg/kg LBM, and 4mg/kg LBM) in central neuropathic pain following spinal cord injury. This arm represents an average of all dextromethorphan doses in combination with 1mg/kg Lidocaine.
- Dextromethorphan/2mg/kg Lidocaine Combination: This randomized, placebo-controlled, double-blind 4x4 factorial crossover clinical trial was part of a larger NIH-funded study to evaluate the analgesic efficacy of multiple dose-combinations of chronic oral (PO)dextromethorphan (placebo, low dose, medium dose, and high dose) and intravenous (IV) lidocaine (0mg/kg LBM, 1mg/kg LBM, 2mg/kg LBM, and 4mg/kg LBM) in central neuropathic pain following spinal cord injury. This arm represents an average of all dextromethorphan doses in combination with 2mg/kg Lidocaine.
- Dextromethorphan/4mg/kg Lidocaine Combination: This randomized, placebo-controlled, double-blind 4x4 factorial crossover clinical trial was part of a larger NIH-funded study to evaluate the analgesic efficacy of multiple dose-combinations of chronic oral (PO)dextromethorphan (placebo, low dose, medium dose, and high dose) and intravenous (IV) lidocaine (0mg/kg LBM, 1mg/kg LBM, 2mg/kg LBM, and 4mg/kg LBM) in central neuropathic pain following spinal cord injury. This arm represents an average of all dextromethorphan doses in combination with 4mg/kg Lidocaine.
Arm/Group | Dextromethorphan/ 0mg/kg Lidocaine Combination | Dextromethorphan/1mg/kg Lidocaine Combination | Dextromethorphan/2mg/kg Lidocaine Combination | Dextromethorphan/4mg/kg Lidocaine Combination
Number analyzed (Participants) | 26 | 26 | 26 | 26
percentage change from baseline | -2.5 (0.0049) | -7.9 (0.0176) | -11.2 (0.0015) | -19.2 (0.0226)
Statistical Analysis 1: Comparison: Dextromethorphan/ 0mg/kg Lidocaine Combination vs Dextromethorphan/1mg/kg Lidocaine Combination vs Dextromethorphan/2mg/kg Lidocaine Combination vs Dextromethorphan/4mg/kg Lidocaine Combination; We performed a lidocaine dose response clinical trial nested within a dextromethorphan clinical trial to evaluate a potential interaction between lidocaine dose and dextromethorphan dose (pain intensity; Gracely scale); Test type: Other — We report the interaction between the lidocaine dose response and dextromethorphan dose response. The type of statistical test was a linear regression model with Chi-square test; p = 0.0322, Pearson's Chi-squared test; Lidocaine dose*dextromethorphan dose = 0.0042, 95% CI 2-sided [0.0004 to 0.0081], Standard Error of Mean 0.0020 — The estimated value is an estimated interaction term, and not a P-value

ADVERSE EVENTS:
Time Frame: Adverse event data were collected from the start of the lidocaine infusion (t=0:00) and recorded for the entire 30 minute infusion (t=0:30)
Groups:
- Placebo Dextromethorphan/0mg/kg Lidocaine Combination; Placebo Dextromethorphan/1mg/kg Lidocaine Combination; Placebo Dextromethorphan/2mg/kg Lidocaine Combination; Placebo Dextromethorphan/4mg/kg Lidocaine Combination; Low Dose Dextromethorphan/0mg/kg Lidocaine Combination; Low Dose Dextromethorphan/1mg/kg Lidocaine Combination; Low Dose Dextromethorphan/2mg/kg Lidocaine Combination; Low Dose Dextromethorphan/4mg/kg Lidocaine Combination; Medium Dose Dextromethorphan/0mg/kg Lidocaine Combination; Medium Dose Dextromethorphan/1mg/kg Lidocaine Combination; Medium Dose Dextromethorphan/2mg/kg Lidocaine Combination; Medium Dose Dextromethorphan/4mg/kg Lidocaine Combination; High Dose Dextromethorphan/0mg/kg Lidocaine Combination; High Dose Dextromethorphan/1mg/kg Lidocaine Combination; High Dose Dextromethorphan/2mg/kg Lidocaine Combination; High Dose Dextromethorphan/4mg/kg Lidocaine Combination: This randomized, placebo-controlled, double-blind 4x4 factorial crossover clinical trial was part of a larger NIH-funded study to evaluate the analgesic efficacy of multiple dose-combinations of chronic oral (PO)dextromethorphan (placebo, low dose, medium dose, and high dose) and intravenous (IV) lidocaine (0mg/kg LBM, 1mg/kg LBM, 2mg/kg LBM, and 4mg/kg LBM) in central neuropathic pain following spinal cord injury.
Arm/Group | Placebo Dextromethorphan/0mg/kg Lidocaine Combination | Placebo Dextromethorphan/1mg/kg Lidocaine Combination | Placebo Dextromethorphan/2mg/kg Lidocaine Combination | Placebo Dextromethorphan/4mg/kg Lidocaine Combination | Low Dose Dextromethorphan/0mg/kg Lidocaine Combination | Low Dose Dextromethorphan/1mg/kg Lidocaine Combination | Low Dose Dextromethorphan/2mg/kg Lidocaine Combination | Low Dose Dextromethorphan/4mg/kg Lidocaine Combination | Medium Dose Dextromethorphan/0mg/kg Lidocaine Combination | Medium Dose Dextromethorphan/1mg/kg Lidocaine Combination | Medium Dose Dextromethorphan/2mg/kg Lidocaine Combination | Medium Dose Dextromethorphan/4mg/kg Lidocaine Combination | High Dose Dextromethorphan/0mg/kg Lidocaine Combination | High Dose Dextromethorphan/1mg/kg Lidocaine Combination | High Dose Dextromethorphan/2mg/kg Lidocaine Combination | High Dose Dextromethorphan/4mg/kg Lidocaine Combination
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/24 | 0/24 | 0/24 | 0/26 | 0/26 | 0/26 | 0/26 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/24 | 0/24 | 0/24 | 0/26 | 0/26 | 0/26 | 0/26 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24 | 0/24
Other Adverse Events (participants affected / at risk) | 4/24 | 3/24 | 5/24 | 10/24 | 5/26 | 7/26 | 8/26 | 15/26 | 3/24 | 6/24 | 6/24 | 15/24 | 3/24 | 3/24 | 6/24 | 17/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo Dextromethorphan/0mg/kg Lidocaine Combination (N=24) | Placebo Dextromethorphan/1mg/kg Lidocaine Combination (N=24) | Placebo Dextromethorphan/2mg/kg Lidocaine Combination (N=24) | Placebo Dextromethorphan/4mg/kg Lidocaine Combination (N=24) | Low Dose Dextromethorphan/0mg/kg Lidocaine Combination (N=26) | Low Dose Dextromethorphan/1mg/kg Lidocaine Combination (N=26) | Low Dose Dextromethorphan/2mg/kg Lidocaine Combination (N=26) | Low Dose Dextromethorphan/4mg/kg Lidocaine Combination (N=26) | Medium Dose Dextromethorphan/0mg/kg Lidocaine Combination (N=24) | Medium Dose Dextromethorphan/1mg/kg Lidocaine Combination (N=24) | Medium Dose Dextromethorphan/2mg/kg Lidocaine Combination (N=24) | Medium Dose Dextromethorphan/4mg/kg Lidocaine Combination (N=24) | High Dose Dextromethorphan/0mg/kg Lidocaine Combination (N=24) | High Dose Dextromethorphan/1mg/kg Lidocaine Combination (N=24) | High Dose Dextromethorphan/2mg/kg Lidocaine Combination (N=24) | High Dose Dextromethorphan/4mg/kg Lidocaine Combination (N=24)
Sedation Complex (Nervous system disorders) | 3 (5) | 3 (7) | 5 (7) | 7 (15) | 5 (7) | 7 (10) | 7 (16) | 14 (36) | 3 (6) | 5 (12) | 4 (8) | 14 (28) | 3 (6) | 2 (2) | 6 (14) | 16 (38) — Dizziness, blurry vision, interference with ability to drive/alertness, etc.
Dry mouth (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 5 (5) | 0 (0) | 0 (0) | 0 (0) | 3 (3) | 2 (2) | 0 (0) | 2 (2) | 4 (4)
Euphoria (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 2 (2)
Parathesias (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 4 (5) | 0 (0) | 2 (3) | 3 (4) | 5 (8) | 0 (0) | 2 (2) | 0 (0) | 7 (8) | 0 (0) | 0 (0) | 2 (3) | 7 (10) — Numbness, tingling, burning
Cramping/Spasms (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No